CLINICAL TRIAL: NCT05937139
Title: The Effect of Breastfeeding Education Given to Fathers Via Whatsapp Messaging Application in the Postpartum Period on Breastfeeding
Brief Title: The Effect of Breastfeeding Education Given to Fathers on Breastfeeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Olcer (Other)
Responsible Party: Sponsor-Investigator, Zeynep Olcer, Assistant Professor, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-81477236-604.01.01-1923
Record Dates: First submitted 2023-06-23; First posted 2023-07-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Breastfeeding
Keywords: breastfeeding; father; training; whatsapp; support
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research is planned to be carried out as an experimental design with four groups of solomon. The randomization of the participants will be made using a computer program and the participants will be assigned to the experimental and control groups in this way
Who Masked: Participant, Care Provider
Masking Description: Participants and the health care provider will not know which group the participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Training group 1 (Experimental): After the scales are applied to the fathers in training group 1 on the 3rd postpartum day, breastfeeding education will begin. The training will last 39 days and the scales will be re-administered on the 42nd postpartum day and at the 12th week postpartum.
  Interventions: Other: Breastfeeding education
- Training group 2 (Experimental): Breastfeeding education will begin to the fathers in training group 2 on the 3rd postpartum day. The training will last 39 days and the scales will be re-administered on the 42nd postpartum day and at the 12th week postpartum.
  Interventions: Other: Breastfeeding education
- Control group 1 (No Intervention): The scales will be administered to the fathers in the control group 2 on the 3rd day, 42nd day, and 12th week postpartum.
- Control group 2 (No Intervention): The scales will be administered to the fathers in the control group 2 on the 42nd day, and 12th week postpartum.

INTERVENTIONS:
Other: Breastfeeding education — Breastfeeding education will be given to fathers.
  Arms: Training group 1; Training group 2

SUMMARY:
The goal of this clinical trial is to determine the effect of breastfeeding education given to fathers via Whatsapp messaging application in the postpartum period on breastfeeding.

The main hypotheses it aims to answer are: ,

* Ho: There is no difference between the "Fathers' Effect on Breastfeeding" scale scores and the Breastfeeding Support Scale scores of the fathers who received breastfeeding training via Whatsapp messaging application in the postpartum period and the scale scores of the fathers who did not receive training.
* H1: There is a difference between the scale scores of the fathers who received breastfeeding training via Whatsapp messaging application in the postpartum period and the scale scores of the fathers who did not receive education.
* H2: There is a difference between the "Breastfeeding Support Scale" scores of fathers who received breastfeeding training via Whatsapp messaging application in the postpartum period and the scale scores of fathers who did not receive education.

Participants will be received breastfeeding training via Whatsapp messaging application in the postpartum period.

If there is a comparison group: Researchers will compare training group and control group to see if effect on breastfeeding.

DETAILED DESCRIPTION:
Spousal and family support increases breastfeeding rates, has a positive effect on the mother-baby relationship, the decisions of mothers who receive emotional support from their spouses are positively affected, women experience less breastfeeding problems when they are consciously supported by their spouses and cope with these problems better, fathers' benefits of breastfeeding It has been reported that the state of knowledge about breastfeeding and its management affects the duration and frequency of breastfeeding. In a study, fathers stated that they wanted to investigate suggestions on how to help their spouses, but there were limited studies on these suggestions so this study was planned .

ELIGIBILITY:
Inclusion Criteria:

* Follow-up of the mother in the postpartum clinic of the hospital
* Feeding the baby with breast milk
* Being an only baby, being at a gestational age of 37 weeks and above, weighing 2500 g and over, not having a congenital disease
* The mother does not have any health problems that may prevent breastfeeding
* The mother and father do not have any barriers to filling out the questionnaire.
* Literacy of mother and father
* Availability of a phone and internet where messages can be read
* Mother and father living in the same house

Exclusion Criteria:

* The baby's inability to get breast milk
* Fathers or mothers have a disability in completing the questionnaire.
* Lack of a phone and internet where messages can be read
* Parents living in separate places

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Support Scale | The scale will be administered to the fathers on the 3rd day postpartum.
  Breastfeeding support of fathers will be evaluated using this scale. Breastfeeding Support Scale is a 5-point Likert-type scale in which the spouses evaluate theirselves' activity while the mother breastfeeding the baby. The lowest score that can be obtained from the scale is 37, and the highest score is 185. A high total score from the whole scale indicates that fathers have a high contribution to breastfeeding.
The Partner Breastfeeding Influence Scale | The scale will be administered to the mothers on the 3rd day postpartum.
  The effect of fathers on breastfeeding will be evaluated with this scale.It is a scale consisting of 14 items and three factors that measures women's social motivations for breastfeeding and spousal support for breastfeeding.Each item that the woman describes as "there is" is given 1 point. The highest score that can be obtained from the scale is 14, and the lowest score is 0. A high score indicates that fathers' support for breastfeeding is high.

SECONDARY OUTCOMES:
Breastfeeding Support Scale | The scale will be administered to the fathers on the 42nd day postpartum.
  Breastfeeding support of fathers will be evaluated using this scale. Breastfeeding Support Scale is a 5-point Likert-type scale in which the spouses evaluate theirselves' activity while the mother breastfeeding the baby. The lowest score that can be obtained from the scale is 37, and the highest score is 185. A high total score from the whole scale indicates that fathers have a high contribution to breastfeeding.
The Partner Breastfeeding Influence Scale | The scale will be administered to the mothers on the 42nd day postpartum.
  The effect of fathers on breastfeeding will be evaluated with this scale.It is a scale consisting of 14 items and three factors that measures women's social motivations for breastfeeding and spousal support for breastfeeding.Each item that the woman describes as "there is" is given 1 point. The highest score that can be obtained from the scale is 14, and the lowest score is 0. A high score indicates that fathers' support for breastfeeding is high.

OTHER OUTCOMES:
Breastfeeding Support Scale | The scale will be administered to the fathers on the 12th week postpartum.
  Breastfeeding support of fathers will be evaluated using this scale. Breastfeeding Support Scale is a 5-point Likert-type scale in which the spouses evaluate theirselves' activity while the mother breastfeeding the baby. The lowest score that can be obtained from the scale is 37, and the highest score is 185. A high total score from the whole scale indicates that fathers have a high contribution to breastfeeding.
The Partner Breastfeeding Influence Scale | The scale will be administered to the mothers on the 12th week postpartum.
  The effect of fathers on breastfeeding will be evaluated with this scale.It is a scale consisting of 14 items and three factors that measures women's social motivations for breastfeeding and spousal support for breastfeeding.Each item that the woman describes as "there is" is given 1 point. The highest score that can be obtained from the scale is 14, and the lowest score is 0. A high score indicates that fathers' support for breastfeeding is high.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep ölçer, Principal Investigator — Ankara Medipol University
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data sets are to be shared IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and any additional supporting information will become available for 1 year after publication
Access Criteria: The data supporting the findings of this studywill be available within the article [and/or] its supplementary materials.

REFERENCES:
- [Result] Bich TH, Hoa DT, Malqvist M. Fathers as supporters for improved exclusive breastfeeding in Viet Nam. Matern Child Health J. 2014 Aug;18(6):1444-53. doi: 10.1007/s10995-013-1384-9. PMID 24162509
- [Result] Moriwaki C, Haku M. Development of a Breastfeeding Support Scale for Couples. J Med Invest. 2016;63(1-2):96-103. doi: 10.2152/jmi.63.96. PMID 27040061
- [Result] Rempel LA, Rempel JK, Moore KCJ. Relationships between types of father breastfeeding support and breastfeeding outcomes. Matern Child Nutr. 2017 Jul;13(3):e12337. doi: 10.1111/mcn.12337. Epub 2016 Jul 27. PMID 27460557